CLINICAL TRIAL: NCT01655550
Title: The Impact of Oral Contrast in Multidetector CT of the Abdomen and Pelvis on Radiologist Confidence: A Randomized Controlled Trial
Brief Title: The Impact of Oral Contrast in Multidetector CT of the Abdomen and Pelvis on Radiologist Confidence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hartford Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GARC003501
Record Dates: First submitted 2012-07-31; First posted 2012-08-02 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-07

CONDITIONS: Routine Outpatients Undergoing Contrast Enhanced CT Scan of the Abdomen and Pelvis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (Other): Patients will get routine CT scans with Oral and Intravenous contrast prior to their CT scan as is routine, standard practice
  Interventions: Other: Withhold oral contrast
- Withold Oral Contrast (Experimental): Subjects will not drink oral contrast, but instead water (in itself a type of contrast agent) prior to their CT. Intravenous contrast will be administered as is routine
  Interventions: Other: Withhold oral contrast

INTERVENTIONS:
Other: Withhold oral contrast — The intervention is to withhold oral contrast

SUMMARY:
The investigators seek to demonstrate the non-superiority of oral contrast versus no oral contrast in intravenously enhanced CT in the outpatient setting. The investigators want to decrease preparation time for the patient and decrease delay in obtaining the study which will ultimately lead to faster results and an increased level of patient convenience.

The investigators hypothesis: Oral contrast does not significantly affect the diagnostic confidence of interpreting radiologists in intravenously enhanced abdominal CT scans.

DETAILED DESCRIPTION:
This study will be a randomized controlled trial comparing radiologist confidence when faced with an intravenously enhanced study with and without oral contrast. At the time of making the appointment, the clerk will ask the patient if he/she wishes to participate in a research study about the impact of oral contrast. If the patient assents, he/she will receive a phone call from a research assistant to obtain informed consent. The first ten patients to call the office to schedule a scan using a 64 slice MDCT will be recruited and randomized if they consent.

Subjects will be randomized at the time of recruitment, which will be when he/she calls to make the appointment for the exam, in a 1:1 ratio between the control arm (contrast) and the experimental arm (no contrast). The control arm will either pick up their two bottles of oral contrast at a radiology office or have the bottles mailed to them as is currently the standard. They will drink the oral contrast two hours before the study. They will also ingest 300 mL of water immediately prior to imaging and be administered the standard intravenous contrast dose. The experimental group will not be mailed or given any oral contrast. They will arrive at their appointment and ingest 300 mL of water immediately prior to the exam as well as the standard intravenous contrast dose and be scanned. This design will eliminate the need to repeat scanning patients, thus decreasing radiation dose. A patient satisfaction survey will be given to each patient following the exam and handed to the technologist

ELIGIBILITY:
Inclusion Criteria:

* order for "Contrast Enhanced abdomen CT" or "Contrast Enhanced abdomen/pelvis CT"

  * age ≥21
  * able and willing to give consent

Exclusion Criteria:

* • allergy to IV contrast

  * order for non-contrast CT
  * <21
  * pregnant woman
  * order for enterography or colonography
  * history of Crohn's Disease or Ulcerative Colitis

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Radiologist Confidence | one-time measurement after scan completion
  Confidence graded by the radiologist on a scale of 1 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M Garcia, MD MHS, Principal Investigator — Hartford Hospital
Locations (1):
- Jefferson Radiology, Hartford, Connecticut, United States